CLINICAL TRIAL: NCT06902493
Title: Impact of Prior Sodium-Glucose Co-Transporter 2 Inhibitor Use on the Development and Progression of Sepsis-Associated Acute Kidney Injury
Brief Title: Impact of Prior SGLT2 Inhibitors Use on the Development and Progression of Sepsis-Associated Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Ahmad Abdullah Salawi, Associate Professor of Pharmaceutics, University of Jazan
Other Study IDs: SGLT2I-AKI
Record Dates: First submitted 2025-03-19; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Sepsis; Septic Shock; Acute Kidney Injury
Keywords: Sepsis; Acute Kidney Injury; Sepsis-associated acute kidney injury; SGLT2i
MeSH Terms: conditions — Sepsis; Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SA-AKI Group: Patients diagnosed with sepsis syndromes (sepsis or septic shock) and AKI according to sepsis-3 definition and KDIGO criteria, respectively
  Interventions: Other: No intervention
- No AKI group: Patients diagnosed with sepsis syndromes (sepsis or septic shock) and AKI according to sepsis-3 definition
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The primary objective of this study is to investigate whether using SGLT2i may be associated with decreased incidence of sepsis-induced AKI or not.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate whether using SGLT2i may be associated with decreased incidence of sepsis-induced AKI or not.

ELIGIBILITY:
Inclusion Criteria:

* All adult (≥ 18 year) patients who were admitted to ICU with sepsis syndromes (sepsis or septic shock), according to sepsis-3 definition.

Exclusion Criteria:

* Missing data
* Renal transplant or tumor
* Solitary kidney
* Established CKD
* Obstructive uropathy
* Renal artery stenosis
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult (≥ 18 year) patients who were admitted to ICU with sepsis syndromes (sepsis or septic shock), according to sepsis-3 definition.
Sampling Method: Probability Sample
Enrollment: 664 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Odds of sepsis-associated acute kidney injury (AKI) in patients with prior use of SGLT2 inhibitors (SGLT2i) | The exposure window for SGLT2i use will be defined as any use within 90 days prior to the onset of sepsis. The outcome (sepsis-associated AKI) will be evaluated during the index hospitalization for sepsis.
  The primary outcome is to determine whether prior use of SGLT2 inhibitors is associated with a reduced odds of developing sepsis-associated AKI. This will be assessed by comparing the frequency of AKI among patients with sepsis who were exposed to SGLT2i prior to hospitalization (cases) versus those who were not exposed (controls).

SECONDARY OUTCOMES:
ICU length of stay | During ICU stay (from ICU admission to discharge), Maximum 6 months stay
  The number of days of ICU stay
The need for RRT | During ICU stay (from ICU admission to discharge), Maximum 6 months stay
  The prevalence of RRT during ICU stay
28-day mortality | Up to day-28 from ICU admission
  The mortality rate at day 28 in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Alshrahili, MSc, Principal Investigator — Armed Forces Hospitals, Southern Region, Saudi Arabia
Locations (1):
- King Fahd Central Hospital, Al ‘Usaylah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No